CLINICAL TRIAL: NCT02589990
Title: Effect of Maximal Strength Training in Relation to Age and Genes
Brief Title: Strength Training Adaptations, Age and Genes
Acronym: STAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South-Eastern Norway (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: STAGE
Record Dates: First submitted 2015-09-24; First posted 2015-10-28 (Estimated); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Healthy
Keywords: health; muscle strength; exercise genomics
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Strength training (Experimental): Strength training, 4 rep of 4RM x 4 sets in leg press.
  Interventions: Behavioral: Strength training

INTERVENTIONS:
Behavioral: Strength training — see arm description

SUMMARY:
The study investigates the effect of maximal strength training on muscular strength and power in different age groups from 20 to 80 year old. It also relates the training adaptations to different known genes such as angiotensin I-converting enzyme (ACE) and Alpha-actinin-3 (ACTN3). Participants will complete an eight weeks, three times per week training intervention of maximal strength training with a pre-post design. In addition, blood samples will be collected for the analyses of genetic variances.

DETAILED DESCRIPTION:
Aim: The study aims to investigate the effect of age and genes on training adaptations to a maximal strength training intervention.

Methods: Participants will be recruited through invitations at work places and other community arenas. The investigators aim to recruit 10-15 subjects in each of the following age groups: 20-29, 30-39, 40-49, 50-59, 60-69 and 70-80 years of age. Both genders will be included. All age groups will be matched for age-related baseline maximal strength and distribution between the two genders. All participants will be checked via a health registration scheme, and excluded if contra indications for hard physical training or testing should appear. When in doubt, the projects physician will decide on inclusion or exclusion due to a thorough examination. Subjects will give a blood sample to be analyzed for known genes such as ACE and ACTN3. The intervention has a pre- post design. Tests of maximal strength and power will be conducted in a leg-press machine, using the protocol assessing one repetition maximum (1RM) previously described. Force and Power will be measured by the Muscle Lab system from Ergotest Tech. (Langesund, Norway). The intervention is an eight week, three times per week protocol, each training session consisting of a standardized warm-up, and 4 repetitions x 4 sets with an intensity of 4 repetition maximum (4RM) performed in the leg press machine.There will be a three minutes pause between sets. Participants will be given instructions and supervision.

Hypothesis: Maximal strength training adaptations will be affected by age and baseline maximal strength but not by gender or genetic variations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 20 to 90 years old

Exclusion Criteria:

* Contraindications to maximum strength training and testing

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2016-01; Primary Completion 2018-08 (Actual); Study Completion 2018-09-03 (Actual)

PRIMARY OUTCOMES:
Maximal muscle strength measured by 1 RM leg press in leg press machine | 8 weeks

SECONDARY OUTCOMES:
Blood sample will be collected to assess gene types Alpha Actinin 3, Angiotensin Converting Enzyme, Angiotensinogen | 8 weeks
rate of force development in leg press measured by MuscleLab (Ergotest Tech., Langesund Norway) | 8 weeks
agility will be measured by counter movement jump using the MuscleLab system by Ergotest Tech. (Langesund, Norway) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Øyvind Støren, PhD, Study Chair — University of South-Eastern Norway; Mona Sæbø, PhD, Study Director — University of South-Eastern Norway
Locations (2):
- Norway (2):
  - Telemark University College, Bø, Telemark
  - Norwegian University of Science and Technology, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Storen O, Helgerud J, Stoa EM, Hoff J. Maximal strength training improves running economy in distance runners. Med Sci Sports Exerc. 2008 Jun;40(6):1087-92. doi: 10.1249/MSS.0b013e318168da2f. PMID 18460997
- [Background] Sunde A, Storen O, Bjerkaas M, Larsen MH, Hoff J, Helgerud J. Maximal strength training improves cycling economy in competitive cyclists. J Strength Cond Res. 2010 Aug;24(8):2157-65. doi: 10.1519/JSC.0b013e3181aeb16a. PMID 19855311